CLINICAL TRIAL: NCT05549466
Title: Antiangiogenic Therapy or Chemotherapy Combined With PD-1 Inhibitor Versus Standard Chemotherapy for PD-1 Inhibitor Refractory R/M NPC
Brief Title: Targeted or Chemotherapy Combined With Immunotherapy Versus Chemotherapy for PD-1 Inhibitor Refractory R/M NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2022-0917
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib; camrelizumab; Drug Therapy; Gemcitabine; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Apatinib plus Camrelizumab and Chemotherapy (Experimental)
  Interventions: Drug: Apatinib, Camrelizumab, Chemotherapy (gemcitabine/ capecitabine/ docetaxel)
- Apatinib plus Camrelizumab (Experimental)
  Interventions: Drug: Apatinib, Camrelizumab
- Camrelizumab and Chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab, Chemotherapy (gemcitabine/ capecitabine/ docetaxel)
- Chemotherapy (Active Comparator)
  Interventions: Drug: Chemotherapy (gemcitabine/ capecitabine/ docetaxel)

INTERVENTIONS:
Drug: Apatinib, Camrelizumab, Chemotherapy (gemcitabine/ capecitabine/ docetaxel) — Gemcitabine, iv, 1000 mg/m^2, D1+D8, Q3W, 6 cycles; or capecitabine, po, 1250 mg/^2, D1-14, BID, Q3W; or docetaxel, iv, 75 mg/m^2, D1, Q3W.
  Apatinib, po, 250mg, qd. Camrelizumab, iv, 200mg, D1, Q3W.
  Arms: Apatinib plus Camrelizumab and Chemotherapy
Drug: Apatinib, Camrelizumab — Apatinib, po, 250mg, qd. Camrelizumab, iv, 200mg, D1, Q3W.
  Arms: Apatinib plus Camrelizumab
Drug: Camrelizumab, Chemotherapy (gemcitabine/ capecitabine/ docetaxel) — Gemcitabine, iv, 1000 mg/m^2, D1+D8, Q3W, 6 cycles; or capecitabine, po, 1250 mg/^2, D1-14, BID, Q3W; or docetaxel, iv, 75 mg/m^2, D1, Q3W.
  Camrelizumab, iv, 200mg, D1, Q3W.
  Arms: Camrelizumab and Chemotherapy
Drug: Chemotherapy (gemcitabine/ capecitabine/ docetaxel) — Gemcitabine, iv, 1000 mg/m^2, D1+D8, Q3W, 6 cycles; or capecitabine, po, 1250 mg/^2, D1-14, BID, Q3W; or docetaxel, iv, 75 mg/m^2, D1, Q3W.
  Arms: Chemotherapy

SUMMARY:
Because most patients with R/M NPC have received long-term maintenance of immunotherapy at the time of initial treatment and the first-line treatment, there are a large number of PD-1 inhibitor refractory patients. How to deal with the ICIs resistance is an urgent problem in clinical practice. Based on previous clinical trials, anti-angiogenic drugs combined with immunotherapy were found to be effective. Therefore, this study intends to preliminarily evaluate which treatment regimen can provide the most benefit to PD-1 inhibitor refractory patients by comparing the efficacy of VEGFR inhibitor or standard chemotherapy combined with PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age;
2. Had histopathologically confirmed nonkeratinizing recurrent/metastatic NPC (AJCC, 8th; the metastatic tissue biopsy is preferred, not necessary).
3. ECOG performance status of 0 or 1.
4. Progression after previous treatment with platinum-based dual-drug chemotherapy.
5. Progression after previous treatment with PD-1 inhibitors.
6. Experieced at least 1 line systemic therapy.
7. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
8. Adequate organ function assessed by laboratory parameters during the screening period
9. Life expectancy more than 12 weeks.
10. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Recurrent lesions suitable for radical treatment (radiotherapy or surgery).
2. Previous treatment over 2 lines.
3. Patients who had previously received one of the three chemotherapy drugs and were randomly assigned to single-agent chemotherapy (control group) were not eligible to reuse the same treatment in this study. In addition, patients who had previously received all three chemotherapy agents for R/M lesions were excluded from the study.
4. Prior use of any anti-VEGF(R) agents.
5. Patients with other malignancies.
6. Patients with nasopharyngeal necrosis found by endoscope before enrollment or with a > 50% chance of nasopharyngeal necrosis according to the risk prediction model: ① Patients with recurrent stage T3-4 received two courses of radiotherapy before enrollment, or received nasopharyngeal radiotherapy within 1 year before enrollment; ② Patients with recurrent T1-2 stage had received two courses of radiotherapy and nasopharyngeal radiotherapy within 1 year before enrollment.
7. Patients with or previous with serious hemorrhage (bleeding >30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).
8. Patients with hypertension who cannot be reduced to the normal range by antihypertensive drug treatment (systolic blood pressure > 140 mmHg/diastolic blood pressure > 90 mmHg), patients with ≥ grade II coronary heart disease, arrhythmia (including QTc interval prolongation > 450 ms in men and > 470 ms in women) and cardiac insufficiency.
9. Patients with known or suspected autoimmune diseases including dementia and seizures.
10. Multiple factors affecting the absorption of oral medications (e.g., dysphagia, chronic diarrhea, and bowel obstruction).
11. An excessive dose of glucocorticoids given within 4 weeks before enrollment.
12. Complications requiring long-term use of immunosuppressive drugs or systemic or local use of immunosuppressive-dose corticosteroids.
13. Patients with active pulmonary tuberculosis (TB) receiving anti-TB treatment or who have received anti-TB treatment within 1 year prior to screening.
14. HIV positive; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C with blood screening positive (HCV antibody positive).
15. Any anti-infective vaccines such as influenza vaccine, varicella vaccine, etc., within 4 weeks before enrollment.
16. Women of childbearing age with a positive pregnancy test and lactating women.
17. Special attention: Patients with active bleeding, ulcers, and bowel perforations within 30 days after major surgery with tumors in close proximity to the internal carotid artery or other major vessels, and those at risk of major bleeding are prohibited.
18. Patients considered unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Objective response rate is the rate of patients achieving complete response or partial response for a certain period of time after intervention.

SECONDARY OUTCOMES:
Median progression-free survival (PFS) | 3 years
  Progression-free survival is calculated from the date of randomization to the date of death of any cause or the first progress at any site, censored on the last date of tumor evaluation if no progress has happened.
Median overall survival (OS) | 3 years
  Overall survival is calculated from the date of randomization to the date of death of any cause, censored on the last date of known survival if no death has happened.
Duration of response (DoR) | 3 years
  Defined as the time from first documentation of objective response to radiological disease progression.
Disease control rate (DCR) | 1 year
  Disease control rate is the rate of patients achieving complete response, partial response or stable disease for at least 4 weeks after intervention.
Adverse events | 3 years
  NCI-CTC5.0 and RTOG standards are adopted, and acute subjective toxicity, acute objective toxicity and late subjective toxicity are included.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-yuan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China